CLINICAL TRIAL: NCT06742801
Title: PELE IDE Clinical Study, Peripheral Onyx™ Liquid Embolic Safety and Effectiveness of The Onyx™ LES for Embolization of Arterial Hemorrhage in the Peripheral Vasculature
Brief Title: Onyx™ Liquid Embolic IDE Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT21044
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Peripheral Arterial Hemorrhage; Trauma; GI Bleed; Ulcer; Hemorrhage
Keywords: Peripheral Arterial Hemorrhage; Embolization treatment
MeSH Terms: conditions — Wounds and Injuries; Gastrointestinal Hemorrhage; Ulcer; Hemorrhage | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment with Onyx LES (Experimental): Device; embolization with liquid embolic
  Interventions: Device: Onyx™ Liquid Embolic System

INTERVENTIONS:
Device: Onyx™ Liquid Embolic System — The proposed indication for Onyx™ LES is: Onyx™ LES is indicated for the embolization of arterial hemorrhage in the peripheral vasculature.
  Other Names: Embolization

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of Onyx™ LES in the treatment of subjects with active arterial bleeding in the peripheral vasculature outside of the heart and brain.

DETAILED DESCRIPTION:
This is a pivotal, prospective, multi-center, non-randomized, single arm study. This study will enroll patients with active arterial bleeding in the peripheral vasculature confirmed by radiologic and/or endoscopic imaging and deemed suitable for embolization treatment by investigator. In this study, peripheral vasculature is defined as outside of the brain and heart.

Up to 135 subjects will be consented to achieve 119 enrolled at up to 25 sites in the US.

This study will have two visits post-index procedure including hospital discharge visit and 30-day follow-up visit. Reintervention visits will be captured through 30 days post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 22 years old.
2. Active arterial bleeding in the peripheral vasculature confirmed by radiologic and/or endoscopic imaging and deemed suitable for embolization treatment by the investigator.

   In this study, peripheral vasculature is defined as outside the brain and heart.
3. Patient or legally authorized representative (LAR) is able to provide written consent to participate in the study.
4. Life expectancy of >30 days, in the opinion of the investigator at the time of enrollment.
5. Target treatment area is free from prior embolization treatment.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Symptoms of active infection.
3. Patient is known to be participating in the study of an investigational drug, biologic, or device.
4. Contrast allergy or other contraindication to angiography, CT, or catheterization, including contrast sensitivity that cannot be adequately treated prior to index procedure.
5. Known allergy to components of Onyx™.
6. Target vasculature unsuitable for the delivery of Onyx™ based upon physician assessment.
7. More than 4 target lesions will require embolization, in the investigator's opinion after imaging-based assessment.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from Arterial Hemorrhage | Through 30 days post-index procedure
  Freedom from arterial hemorrhage in all target location(s) after treatment with Onyx™ LES at the index procedure without re-embolization or any other intervention at the target location(s) due to persistent or recurrent hemorrhage through 30 days. Freedom from arterial hemorrhage where an arterial hemorrhage event is defined as a type 3 or greater BARC bleeding criteria as assessed by the Clinical Events Committee (CEC) through 30 days.
Freedom from System-related Major Adverse Events (MAE) | Through 30 days post-index procedure
  The primary safety endpoint is defined as freedom from system-related Major Adverse Events (MAE) through 30 days after the point of enrollment as assessed by the CEC.

SECONDARY OUTCOMES:
Procedural Success | At the completion of the index procedure
  successful delivery and deployment of Onyx™ to the target location without non-target embolization or Onyx™ cast migration and the successful removal of the delivery system at the completion of the index procedure.
Technical Success | At the completion of the index procedure
  Technical Success is defined as absence of angiographic signs of bleeding after Onyx ™ embolization at each target location based on core lab assessment.
Reintervention | Through 30 days post-index procedure
  Reintervention is defined as the number of additional procedures needed to treat the target location(s) embolized with Onyx™ through 30 days following the index procedure.
Transfusions | Through 30 days post-index procedure
  Transfusions defined as the number of blood transfusions required post-index procedure through 30 days will use blood transfusions starting after the removal of the delivery system. The number of blood units used for each transfusion will also be collected.

OTHER OUTCOMES:
Ancillary Endpoint | Through index procedure
  Duration of the index procedure
Ancillary Endpoint | Through 30 days post-index procedure
  Length of hospitalization, post-index procedure
Ancillary Endpoint | Through 30 days post-index procedure
  Tabulate adjunctive use of other types of embolic agents to treat target locations at index procedure and reinterventions

CONTACTS AND LOCATIONS:
Overall Officials: Osman Ahmed, MD, Principal Investigator — University of Chicago
Locations (13):
- United States (13):
  - Mayo Clinic, Phoenix, Arizona
  - University of California, Irvine, Irvine, California
  - Stanford Medical Center, Palo Alto, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Yale New Haven, New Haven, Connecticut
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Masschusetts General Hospital, Boston, Massachusetts
  - CHI Health Creighton University Medical Center-Bergan-Mercy, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - The Mount Sinai, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Univ Of Texas Southwestern, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No